CLINICAL TRIAL: NCT03447236
Title: An Evaluation of Changes in Brain Functional Connectivity Resulting From Cognitive Intervention by Means of the Feuerstein Instrumental Enrichment Program in Older People With Mild Cognitive Impairment (MCI)
Brief Title: Functional MRI Changes Resulting From the Feuerstein Program in Older People With Mild Cognitive Impairment (MCI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Adolf und Mary Mil-Stiftung (Other); Helen Bader Foundation (Unknown); Montreal Jewish Community Fund (Unknown); Rochlin Family Foundation (Unknown)
Responsible Party: Principal Investigator, Tzvi Dwolatzky, Director Geriatrics, Rambam Health Care Campus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0580-16-RMB
Record Dates: First submitted 2018-02-18; First posted 2018-02-27 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Mild Cognitive Impairment
Keywords: Older people; Cognitive training; MCI
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Feuerstein Program (Experimental): All subjects participating in the Feuerstein Program will be evaluated by anatomical and functional MRI as well as computerized cognitive assessment prior to and following intervention as outlined in the protocol.
  Interventions: Behavioral: Feuerstein Program

INTERVENTIONS:
Behavioral: Feuerstein Program — Mediated learning cognitive enhancement program

SUMMARY:
Background: The Feuerstein Instrumental Enrichment Program was designed to prevent mental deterioration and preserve cognitive abilities among people aged 60 and above. The program is an applied practicable program based on the theories of Structural Cognitive Modifiability as well as on a Mediated Learning Experience. The program takes into consideration the unique characteristics and requirements of the older population. The program is composed of a variety of cognitive tasks that offer systematic activities intended to stimulate mental and cognitive development.

Objective: To examine the influence of the Feuerstein Program on brain functional connectivity as measured by MRI assessments and cognitive function of participants suffering from Mild Cognitive Impairment (MCI).

Hypothesis: The Feuerstein Program will improve cognitive abilities and affect brain functional connectivity.

Methods: Residents of retirement homes will be offered to participate in the study. Participants will undergo cognitive and MRI assessments prior to and following a period of cognitive intervention using the Feuerstein Instrumental Enrichment Program.

DETAILED DESCRIPTION:
Introduction

In recent decades, with the increase in life expectancy, the number of older people and their relative rate within the population have risen dramatically. This trend led to increased rates of people suffering from a mild cognitive disorder and dementia in developed countries. Mild Neurocognitive Disorder or Mild Cognitive Impairment (MCI) is defined as a transition state between successful aging and a state of dementia. This state is characterized by cognitive impairment and a decline in memory skills while daily functioning is maintained.

Older people diagnosed with MCI are at increased risk of developing dementia, particularly Alzheimer's disease. This risk is ranked at about 12% every year.

Since this is a pre-dementia stage, great importance lies in finding methods that may prevent or at least decelerate the progress of MCI to dementia. Cognitive training is believed to be an appropriate intervention for preserving cognitive function.

The Feuerstein Program

This program is designed to prevent mental deterioration and preserve cognitive abilities among people aged 60 and above (hereinafter "The Feuerstein Program"). The program is the initiative and brainchild of Professor Reuven Feuerstein - Israel Prize Laureate, founder and President of the Feuerstein Institute for the Enhancement of Learning Potential.

The program is based on the theories of Structural Cognitive Modifiability as well as on Mediated Learning Experience. For the needs of this program, the tools were suited to the unique characteristics and requirements of the older population.

The program is composed of a variety of tools (hereinafter: instrumental enrichment) that offer systematic activities intended to stimulate mental and cognitive development.

Instrumental enrichment is a set of tools dealing with required thinking skills to promote learning and thinking processes. The tasks of the various tools are free of educational content and they engage in pure learning and thinking processes. The tools are delivered through a special mediation approach, in which teachers and supervisors are trained in specialized courses.

Objectives of the Feuerstein Program

The main objective: to enhance the transformation (variability) capacity of a human being.

The sub-objectives:

1. Correction and development of defective thinking skills, that are responsible for learning difficulties and the absence of transformation (variability).
2. Equipping the learner with literal and conceptual content that he requires during his learning processes.
3. Creating and establishing proper sound thinking and working habits.
4. Creating insight and awareness regarding the processes involved in learning.
5. Creating internal motivation for carrying out tasks.

The Learning Process

The instrumental enrichment tools are distributed to the participant as work sheets. The teacher creates a "mediating" dialogue between himself and the participants, thus enabling them to construct learning skills and essential thinking strategies. In addition, the teacher bridges the learning skills that were studied to the daily life of the older participant.

Products

1. Creating within them awareness to their learning and thinking processes (Metacognition) while introducing an optimistic and positive attitude towards the ability to effect a significant change in these areas.
2. Instill the older person with control over his thinking skills.
3. Enhancing the sense of capability of the older person.

The Intervention Focuses of the Instrumental Enrichment Tools that will be utilized in the Program

1. Methodical information gathering.
2. Orientation and function in space and time.
3. Comparison and sorting capabilities.
4. Memory.
5. Raising hypotheses and their examination.
6. Perspicuousness (clear wording) and naming capabilities.

MRI imaging

The current study includes anatomical and functional MRI imaging in order to evaluate the relationship between cognitive changes and brain functional connectivity.

Research Objective

Examining the effects of the Feuerstein Program on brain functional connectivity as measured by MRI and cognitive function assessed by a computerized cognitive battery in subjects with MCI.

Research Hypothesis

The Feuerstein Program will improve cognitive abilities and affect brain functional connectivity.

Methodology

An open-label single group interventional study.

Research Assessment Tools

1. Cognitive screening by means of the MoCA (Montreal Cognitive Assessment) Test.
2. CogSym (Cognitive Symptom) Meta-cognition questionnaire composed of ten items related to the cognitive ability of the examinee during his daily functioning. The examinee is asked to assess for each item, what is his ability level for the function being described, on a 5 levels scale (1 = excellent, 5 = inferior).
3. World Health Organization well-being index questionnaire.
4. The Neurotrax computerized cognitive assessment battery.
5. Anatomical and functional MRI imaging

The intervention

Phase 1:

15 participants will undergo the aforementioned assessments at baseline followed by an intervention period involving 30 twice weekly sessions of the Feuerstein Program each lasting 90 minutes over 15 weeks. Assessments will be repeated after session 30 and finally at 9 months following intervention commencement.

Phase 2:

15 participants will undergo the aforementioned assessments initially, followed by a waiting period of 15 weeks without intervention (baseline function). This will be followed by an intervention period involving 30 twice weekly sessions of the Feuerstein Program each lasting 90 minutes over 15 weeks. Assessments will be repeated after session 30 and finally at 9 months following intervention commencement.

Data Analysis The statistical analysis will be conducted as is customary in clinical research within the field.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 60 and above.
2. Hebrew speakers.
3. Expressing willingness to participate in the research and deliberately signing a consent form.
4. A diagnosis of MCI exists according to accepted clinical criteria - the examinee's score in the MoCA Test is within the range of 18-26 (inclusive).

Exclusion Criteria:

1. A medical or functional condition that will not allow the subject to participate in the intervention program within the research period.
2. Diagnosed subjects suffering from active depression, bipolar disorder or schizophrenia.
3. Subjects who suffer from a diagnosed cognitive impairment other than MCI (delirium dementia or mental retardation).
4. Visual impairment that will not allow subjects to observe detailed information on a 32' screen from a distance of 1 meter.
5. Hearing impairment that will not allow subjects to listen to instructions during assessment.
6. Subjects whose MoCA Test's score is 17 and below or 27 and above.
7. Subjects unable to undergo MRI assessments based on a standard questionnaire of eligibility for MRI excluding the use of metal and electronic implants.
8. Subjects who will decide not to participate following a 10 minute MRI scan which will allow subjects to experience the procedure.
9. The finding of a Random Space Occupying Lesion on MRI scan at initial anatomical assessment.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-07-04 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline functional connectivity | Through study completion, an average of 11 months
  Based on correlation coefficient of FMRI signal between brain regions

SECONDARY OUTCOMES:
Change from baseline cognitive function | Through study completion, an average of 11 months
  Based on Neurotrax computerized neuropsychological assessment battery

CONTACTS AND LOCATIONS:
Overall Officials: Tzvi Dwolatzky, MD MBBCh, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dwolatzky T, Whitehead V, Doniger GM, Simon ES, Schweiger A, Jaffe D, Chertkow H. Validity of a novel computerized cognitive battery for mild cognitive impairment. BMC Geriatr. 2003 Nov 2;3:4. doi: 10.1186/1471-2318-3-4. PMID 14594456
- [Background] Lifshitz M, Dwolatzky T, Press Y. Validation of the Hebrew version of the MoCA test as a screening instrument for the early detection of mild cognitive impairment in elderly individuals. J Geriatr Psychiatry Neurol. 2012 Sep;25(3):155-61. doi: 10.1177/0891988712457047. PMID 23124009
- [Background] Hostage CA, Choudhury KR, Murali Doraiswamy P, Petrella JR; Alzheimer's Disease Neuroimaging Initiative. Mapping the effect of the apolipoprotein E genotype on 4-year atrophy rates in an Alzheimer disease-related brain network. Radiology. 2014 Apr;271(1):211-9. doi: 10.1148/radiol.13131041. Epub 2013 Dec 12. PMID 24475827
- [Background] Esposito R, Mosca A, Pieramico V, Cieri F, Cera N, Sensi SL. Characterization of resting state activity in MCI individuals. PeerJ. 2013 Aug 20;1:e135. doi: 10.7717/peerj.135. eCollection 2013. PMID 24010015
- [Background] Deng Y, Liu K, Shi L, Lei Y, Liang P, Li K, Chu WC, Wang D; Alzheimer's Disease Neuroimaging Initiative. Identifying the Alteration Patterns of Brain Functional Connectivity in Progressive Mild Cognitive Impairment Patients: A Longitudinal Whole-Brain Voxel-Wise Degree Analysis. Front Aging Neurosci. 2016 Aug 17;8:195. doi: 10.3389/fnagi.2016.00195. eCollection 2016. PMID 27582703
- [Background] Li Y, Wang X, Li Y, Sun Y, Sheng C, Li H, Li X, Yu Y, Chen G, Hu X, Jing B, Wang D, Li K, Jessen F, Xia M, Han Y. Abnormal Resting-State Functional Connectivity Strength in Mild Cognitive Impairment and Its Conversion to Alzheimer's Disease. Neural Plast. 2016;2016:4680972. doi: 10.1155/2016/4680972. Epub 2015 Dec 30. PMID 26843991
- [Background] Meskaldji DE, Preti MG, Bolton TA, Montandon ML, Rodriguez C, Morgenthaler S, Giannakopoulos P, Haller S, Van De Ville D. Prediction of long-term memory scores in MCI based on resting-state fMRI. Neuroimage Clin. 2016 Oct 11;12:785-795. doi: 10.1016/j.nicl.2016.10.004. eCollection 2016. PMID 27812505
- [Background] Wells RE, Yeh GY, Kerr CE, Wolkin J, Davis RB, Tan Y, Spaeth R, Wall RB, Walsh J, Kaptchuk TJ, Press D, Phillips RS, Kong J. Meditation's impact on default mode network and hippocampus in mild cognitive impairment: a pilot study. Neurosci Lett. 2013 Nov 27;556:15-9. doi: 10.1016/j.neulet.2013.10.001. Epub 2013 Oct 10. PMID 24120430
- [Background] Eyre HA, Acevedo B, Yang H, Siddarth P, Van Dyk K, Ercoli L, Leaver AM, Cyr NS, Narr K, Baune BT, Khalsa DS, Lavretsky H. Changes in Neural Connectivity and Memory Following a Yoga Intervention for Older Adults: A Pilot Study. J Alzheimers Dis. 2016;52(2):673-84. doi: 10.3233/JAD-150653. PMID 27060939
- [Background] Topp CW, Ostergaard SD, Sondergaard S, Bech P. The WHO-5 Well-Being Index: a systematic review of the literature. Psychother Psychosom. 2015;84(3):167-76. doi: 10.1159/000376585. Epub 2015 Mar 28. PMID 25831962
- [Background] Karahanoglu FI, Van De Ville D. Transient brain activity disentangles fMRI resting-state dynamics in terms of spatially and temporally overlapping networks. Nat Commun. 2015 Jul 16;6:7751. doi: 10.1038/ncomms8751. PMID 26178017
- [Background] Allan TW, Francis ST, Caballero-Gaudes C, Morris PG, Liddle EB, Liddle PF, Brookes MJ, Gowland PA. Functional Connectivity in MRI Is Driven by Spontaneous BOLD Events. PLoS One. 2015 Apr 29;10(4):e0124577. doi: 10.1371/journal.pone.0124577. eCollection 2015. PMID 25922945